CLINICAL TRIAL: NCT00459017
Title: The Effect of Frequent Self Measurements of Blood Pressure on the Control of Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA -02-2773-YM-CTIL
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Hypertension
Keywords: 24 hour ambulatory blood pressure measurement; Mean blood pressure; Wrist manometer; Frequent measurement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Portable blood pressure wrist manometer

SUMMARY:
Despite knowledge regarding the importance of controlling patients' blood pressure (BP) only 30% of treated patients achieve BP goals. Our objective was to determine the effect of frequent self measurements of BP in the patients' natural environment as a mean to improve BP control. Our hypothesis was that frequent measurements of BP will reduce mean BP levels.

ELIGIBILITY:
Inclusion Criteria:

* Signing an informed consent form
* Having a diagnosis of hypertension for more than one year according to patients'records.
* receiving at least one medication for hypertension
* A reasonable understanding of Hebrew
* An ambulatory state enabling regular visits to a primary physician in the community and self-measurement of hypertension using the electronic device

Exclusion Criteria:

* Lack of willingness to participate in the study.Known arrhythmia
* Malignant disease
* Poor understanding of Hebrew

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-12; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Meam blood pressure

SECONDARY OUTCOMES:
Satisfaction
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Maor, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Kupat Holim Meuhedet, Tel Aviv, Israel